CLINICAL TRIAL: NCT04884945
Title: Pediatric Robotic Versus Open Pyeloplasty: A Pilot Randomized Control Study
Brief Title: Pediatric Robotic Versus Open Pyeloplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to resume recruitment post COVID.
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Benjamin Whittam, Associate Professor Urology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1403886306
Record Dates: First submitted 2020-11-10; First posted 2021-05-13 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Urology; Ureteropelvic Junction Obstruction
Keywords: patient centered outcomes
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Intervention Model Description: For Aim 2: For the RCT, patients are randomized to either RALP or OP by using a pool of 20 cards of which 10 say "robotic surgery" and 10 say "open surgery.
Who Masked: Participant, Care Provider
Masking Description: Patient, Family, and Nursing Staff on Surgical Floor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Robotic Surgery (Active Comparator): Robotic-Assisted Laparoscopic Pyeloplasty (RALP), standard of care treatment option for UPJ obstruction
  Interventions: Device: Robotic-Assisted Laparoscopic Pyeloplasty (RALP)
- Open Surgery (Active Comparator): Open Pyeloplasty (OP), standard of care treatment option for UPJ obstruction
  Interventions: Procedure: Open Pyeloplasty (OP)

INTERVENTIONS:
Procedure: Open Pyeloplasty (OP) — Open approach for the surgical correction of UPJ obstruction
  Arms: Open Surgery
Device: Robotic-Assisted Laparoscopic Pyeloplasty (RALP) — Robotic approach with the da Vinci Surgical System for the surgical correction of UPJ obstruction
  Arms: Robotic Surgery

SUMMARY:
The objective is conduct a pilot randomized controlled trial comparing robotic and open techniques for surgical correction of congenital UPJ obstruction (pyeloplasty) in pediatric patients. This study will serve as a proof of concept trial to demonstrate feasibility of recruiting pediatric patients to participate in a randomized study for surgical procedures and delineate patient-centered outcomes. Should this study prove randomization is feasible, a randomized comparative effectiveness trial with sufficient power to determine whether open or robotic-assisted pyeloplasty has superior patient-centered outcomes will be pursued.

DETAILED DESCRIPTION:
Technological innovations are an ongoing reality in clinical medicine, most dramatically in the operating room. Each advance is often heralded as an improvement in patient care, promising to correct deficiencies and advance standard operative procedures. Unfortunately, these new technologies often lack sufficient evidence to support such claims. Robotic assisted laparoscopic (RAL) surgery continues to gain popularity among pediatric surgical specialists, particularly for reconstructive procedures such as correction of ureteropelvic junction (UPJ) obstruction or vesicoureteral reflux (VUR).In these operations, where traditional open surgery yields a nearly 95% clinical success rate it is difficult to demonstrate improvement with a new surgical technique. Despite these impressive outcomes with the open approach many pediatric urologists are shifting towards newer RAL approaches, claiming faster recovery and improved cosmesis with a nominal increase in surgical cost.

There is a striking dearth of comparative effectiveness research in pediatric surgical specialties, especially given the wide range of available therapies for a variety of surgical problems. Conducting randomized controlled trials of surgical interventions can be very difficult, especially in the pediatric population.

Currently, all studies of pediatric robotic surgery have focused on traditional outcomes, e.g., length of stay, pain scores, pain medication usage, scar perception, cost analysis, and capital gains benefits. While these measures are important to study, the investigators believe that researchers must also focus on patients' treatment experiences or patients' evaluations of their own outcomes. By focusing on these 'patient-centered outcomes' the investigators will be able to improve outcomes from surgical procedures in ways that are most important to patients and their families.

We propose a pilot randomized controlled trial comparing robotic and open techniques for surgical correction of congenital UPJ obstruction (pyeloplasty) in pediatric patients. This study will serve as a proof of concept trial to demonstrate feasibility of recruiting pediatric patients to participate in a randomized study for surgical procedures and delineate patient-centered outcomes. Should this study prove randomization is feasible, the investigators will seek funding to conduct a large, randomized comparative effectiveness trial with sufficient power to determine whether open or robotic-assisted pyeloplasty has superior patient-centered outcomes.

The investigators propose to accomplish these goals with the following Specific Aims:

Aim 1: Utilize novel patient-centered research methods to:

* Identify outcomes of importance to patients and families related to pediatric pyeloplasty.
* Determine patient and family preferences regarding acceptability of randomization and blinding of pediatric surgical patients and construct a recruitment approach to achieve enrollment.

Aim 2: Conduct a randomized pilot study with goal of enrolling ten to twenty pediatric patients (age 2 - 8 years) to either open or robotic pyeloplasty for treatment of primary UPJ obstruction.

Sub Aim 2a: Collect preliminary data regarding the patient-centered outcomes identified in Aim 1.

Sub Aim 2b: Evaluate the effectiveness of the recruitment approach for randomized surgical studies developed in Aim 1.

The investigators believe that the use of innovative and novel patient-centered research methods will lead to a significant breakthrough in developing a recruitment approach that is both acceptable to pediatric patients/families and optimizes participant willingness to participate in RCTs of surgical interventions. Additionally these same innovative research methods will allows the investigators to explore what outcomes are meaningful to patients and families, which will hopefully allow the care team to counsel patients and families in a way that maximizes their chances of achieving patient- and family-centered goals.

ELIGIBILITY:
For Aim 2:

Inclusion Criteria:

* Primary UPJ obstruction diagnosed by scan and presenting to the pediatric urology clinic for evaluation
* Patient between age 2 - 8 years old

Exclusion Criteria:

* Serious comorbidities (cardiovascular or respiratory disease, or other congenital anomalies requiring surgical intervention).
* BMI greater than the 95th %tile for age.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Whittam, MD, Principal Investigator — Riley Children's Health, Indiana University Health, Pediatric Urology
Locations (1):
- Riley Children's Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Monn MF, Bahler CD, Schneider EB, Whittam BM, Misseri R, Rink RC, Sundaram CP. Trends in robot-assisted laparoscopic pyeloplasty in pediatric patients. Urology. 2013 Jun;81(6):1336-41. doi: 10.1016/j.urology.2013.01.025. Epub 2013 Mar 19. PMID 23522294
- [Background] Liu DB, Ellimoottil C, Flum AS, Casey JT, Gong EM. Contemporary national comparison of open, laparoscopic, and robotic-assisted laparoscopic pediatric pyeloplasty. J Pediatr Urol. 2014 Aug;10(4):610-5. doi: 10.1016/j.jpurol.2014.06.010. Epub 2014 Jul 11. PMID 25082711
- [Background] Steffens J, Langen PH, Haben B, Hiebl R, Steffens L, Polsky MS. Politano-leadbetter ureteroneocystostomy. A 30-year experience. Urol Int. 2000;65(1):9-14. doi: 10.1159/000064827. PMID 10965295
- [Background] Shaul DB, Cunningham JA, Lowe P, Skaist LB, Hardy BE. Infant pyeloplasty is a low-risk procedure. J Pediatr Surg. 1994 Feb;29(2):343-7. doi: 10.1016/0022-3468(94)90345-x. PMID 8176617
- [Background] Hendren WH, Radhakrishnan J, Middleton AW Jr. Pediatric pyleoplasty. J Pediatr Surg. 1980 Apr;15(2):133-44. doi: 10.1016/s0022-3468(80)80004-2. PMID 7373488
- [Background] Salem YH, Majd M, Rushton HG, Belman AB. Outcome analysis of pediatric pyeloplasty as a function of patient age, presentation and differential renal function. J Urol. 1995 Nov;154(5):1889-93. PMID 7563377
- [Background] Behan JW, Kim SS, Dorey F, De Filippo RE, Chang AY, Hardy BE, Koh CJ. Human capital gains associated with robotic assisted laparoscopic pyeloplasty in children compared to open pyeloplasty. J Urol. 2011 Oct;186(4 Suppl):1663-7. doi: 10.1016/j.juro.2011.04.019. PMID 21862079
- [Background] Lee RS, Retik AB, Borer JG, Peters CA. Pediatric robot assisted laparoscopic dismembered pyeloplasty: comparison with a cohort of open surgery. J Urol. 2006 Feb;175(2):683-7; discussion 687. doi: 10.1016/S0022-5347(05)00183-7. PMID 16407025
- [Background] Cundy TP, Harling L, Hughes-Hallett A, Mayer EK, Najmaldin AS, Athanasiou T, Yang GZ, Darzi A. Meta-analysis of robot-assisted vs conventional laparoscopic and open pyeloplasty in children. BJU Int. 2014 Oct;114(4):582-94. doi: 10.1111/bju.12683. PMID 25383399
- [Background] Barbosa JA, Barayan G, Gridley CM, Sanchez DC, Passerotti CC, Houck CS, Nguyen HT. Parent and patient perceptions of robotic vs open urological surgery scars in children. J Urol. 2013 Jul;190(1):244-50. doi: 10.1016/j.juro.2012.12.060. Epub 2012 Dec 28. PMID 23276511
- [Background] Bennett WE Jr, Whittam BM, Szymanski KM, Rink RC, Cain MP, Carroll AE. Validated cost comparison of open vs. robotic pyeloplasty in American children's hospitals. J Robot Surg. 2017 Jun;11(2):201-206. doi: 10.1007/s11701-016-0645-1. Epub 2016 Oct 20. PMID 27766551
- [Background] Ferreira LM. Surgical randomized controlled trials: reflection of the difficulties. Acta Cirurgica Brasileira 2005;19(Suppl 1):2-3.
- [Background] McCulloch P, Taylor I, Sasako M, Lovett B, Griffin D. Randomised trials in surgery: problems and possible solutions. BMJ. 2002 Jun 15;324(7351):1448-51. doi: 10.1136/bmj.324.7351.1448. No abstract available. PMID 12065273
- [Background] Caldwell PH, Murphy SB, Butow PN, Craig JC. Clinical trials in children. Lancet. 2004 Aug 28-Sep 3;364(9436):803-11. doi: 10.1016/S0140-6736(04)16942-0. PMID 15337409
- [Background] Curry JI, Reeves B, Stringer MD. Randomized controlled trials in pediatric surgery: could we do better? J Pediatr Surg. 2003 Apr;38(4):556-9. doi: 10.1053/jpsu.2003.50121. PMID 12677565
- [Background] Rosenthal R, Kasenda B, Dell-Kuster S, von Elm E, You J, Blumle A, Tomonaga Y, Saccilotto R, Amstutz A, Bengough T, Meerpohl JJ, Stegert M, Tikkinen KA, Neumann I, Carrasco-Labra A, Faulhaber M, Mulla S, Mertz D, Akl EA, Bassler D, Busse JW, Ferreira-Gonzalez I, Lamontagne F, Nordmann A, Gloy V, Olu KK, Raatz H, Moja L, Ebrahim S, Schandelmaier S, Sun X, Vandvik PO, Johnston BC, Walter MA, Burnand B, Schwenkglenks M, Hemkens LG, Bucher HC, Guyatt GH, Briel M. Completion and Publication Rates of Randomized Controlled Trials in Surgery: An Empirical Study. Ann Surg. 2015 Jul;262(1):68-73. doi: 10.1097/SLA.0000000000000810. PMID 24979608
- [Background] Casella DP, Fox JA, Schneck FX, Cannon GM, Ost MC. Cost analysis of pediatric robot-assisted and laparoscopic pyeloplasty. J Urol. 2013 Mar;189(3):1083-6. doi: 10.1016/j.juro.2012.08.259. Epub 2012 Sep 24. PMID 23017518
- [Background] Yu HY, Hevelone ND, Lipsitz SR, Kowalczyk KJ, Hu JC. Use, costs and comparative effectiveness of robotic assisted, laparoscopic and open urological surgery. J Urol. 2012 Apr;187(4):1392-8. doi: 10.1016/j.juro.2011.11.089. Epub 2012 Feb 16. PMID 22341274
- [Background] Cundy TP, Shetty K, Clark J, Chang TP, Sriskandarajah K, Gattas NE, Najmaldin A, Yang GZ, Darzi A. The first decade of robotic surgery in children. J Pediatr Surg. 2013 Apr;48(4):858-65. doi: 10.1016/j.jpedsurg.2013.01.031. PMID 23583146
- [Background] Tanaka ST, Grantham JA, Thomas JC, Adams MC, Brock JW 3rd, Pope JC 4th. A comparison of open vs laparoscopic pediatric pyeloplasty using the pediatric health information system database--do benefits of laparoscopic approach recede at younger ages? J Urol. 2008 Oct;180(4):1479-85. doi: 10.1016/j.juro.2008.06.044. Epub 2008 Aug 16. PMID 18710777
- [Background] Fowler FJ Jr, Barry MJ, Lu-Yao G, Wasson J, Roman A, Wennberg J. Effect of radical prostatectomy for prostate cancer on patient quality of life: results from a Medicare survey. Urology. 1995 Jun;45(6):1007-13; discussion 1013-5. doi: 10.1016/s0090-4295(99)80122-8. PMID 7771002
- [Background] Resnick MJ, Barocas DA, Morgans AK, Phillips SE, Koyama T, Albertsen PC, Cooperberg MR, Goodman M, Greenfield S, Hamilton AS, Hoffman KE, Hoffman RM, Kaplan SH, McCollum D, Paddock LE, Stanford JL, Stroup AM, Wu XC, Penson DF. The Evolution of Self-Reported Urinary and Sexual Dysfunction over the Last Two Decades: Implications for Comparative Effectiveness Research. Eur Urol. 2015 Jun;67(6):1019-1025. doi: 10.1016/j.eururo.2014.08.035. Epub 2014 Aug 28. PMID 25174325
- [Background] Morin L, Cendron M, Crombleholme TM, Garmel SH, Klauber GT, D'Alton ME. Minimal hydronephrosis in the fetus: clinical significance and implications for management. J Urol. 1996 Jun;155(6):2047-9. doi: 10.1016/s0022-5347(01)66102-0. PMID 8618331
- [Background] Persky L, Krause JR, Boltuch RL. Initial complications and late results in dismembered pyeloplasty. J Urol. 1977 Jul;118(1 Pt 2):162-5. doi: 10.1016/s0022-5347(17)57936-7. PMID 875213
- [Background] Psooy K, Pike JG, Leonard MP. Long-term followup of pediatric dismembered pyeloplasty: how long is long enough? J Urol. 2003 May;169(5):1809-12; discussion 1812; author reply 1812. doi: 10.1097/01.ju.0000055040.19568.ea. PMID 12686849
- [Background] Riachy E, Cost NG, Defoor WR, Reddy PP, Minevich EA, Noh PH. Pediatric standard and robot-assisted laparoscopic pyeloplasty: a comparative single institution study. J Urol. 2013 Jan;189(1):283-7. doi: 10.1016/j.juro.2012.09.008. Epub 2012 Nov 20. PMID 23174238
- [Background] Penn HA, Gatti JM, Hoestje SM, DeMarco RT, Snyder CL, Murphy JP. Laparoscopic versus open pyeloplasty in children: preliminary report of a prospective randomized trial. J Urol. 2010 Aug;184(2):690-5. doi: 10.1016/j.juro.2010.03.062. Epub 2010 Jun 19. PMID 20639039
- [Background] Mei H, Pu J, Yang C, Zhang H, Zheng L, Tong Q. Laparoscopic versus open pyeloplasty for ureteropelvic junction obstruction in children: a systematic review and meta-analysis. J Endourol. 2011 May;25(5):727-36. doi: 10.1089/end.2010.0544. Epub 2011 Apr 8. PMID 21476861
- [Background] Piaggio LA, Franc-Guimond J, Noh PH, Wehry M, Figueroa TE, Barthold J, Gonzalez R. Transperitoneal laparoscopic pyeloplasty for primary repair of ureteropelvic junction obstruction in infants and children: comparison with open surgery. J Urol. 2007 Oct;178(4 Pt 2):1579-83. doi: 10.1016/j.juro.2007.03.159. Epub 2007 Aug 16. PMID 17707047
- [Background] Yohannes P, Rotariu P, Pinto P, Smith AD, Lee BR. Comparison of robotic versus laparoscopic skills: is there a difference in the learning curve? Urology. 2002 Jul;60(1):39-45; discussion 45. doi: 10.1016/s0090-4295(02)01717-x. PMID 12100918
- [Background] Lim PC, Kang E, Park DH. A comparative detail analysis of the learning curve and surgical outcome for robotic hysterectomy with lymphadenectomy versus laparoscopic hysterectomy with lymphadenectomy in treatment of endometrial cancer: a case-matched controlled study of the first one hundred twenty two patients. Gynecol Oncol. 2011 Mar;120(3):413-8. doi: 10.1016/j.ygyno.2010.11.034. Epub 2010 Dec 30. PMID 21194735
- [Background] Sorensen MD, Delostrinos C, Johnson MH, Grady RW, Lendvay TS. Comparison of the learning curve and outcomes of robotic assisted pediatric pyeloplasty. J Urol. 2011 Jun;185(6 Suppl):2517-22. doi: 10.1016/j.juro.2011.01.021. Epub 2011 Apr 28. PMID 21555027
- [Background] Chandra V, Nehra D, Parent R, Woo R, Reyes R, Hernandez-Boussard T, Dutta S. A comparison of laparoscopic and robotic assisted suturing performance by experts and novices. Surgery. 2010 Jun;147(6):830-9. doi: 10.1016/j.surg.2009.11.002. Epub 2009 Dec 31. PMID 20045162
- [Background] Varda BK, Johnson EK, Clark C, Chung BI, Nelson CP, Chang SL. National trends of perioperative outcomes and costs for open, laparoscopic and robotic pediatric pyeloplasty. J Urol. 2014 Apr;191(4):1090-5. doi: 10.1016/j.juro.2013.10.077. Epub 2013 Oct 25. PMID 24513164
- [Background] Dangle PP, Kearns J, Anderson B, Gundeti MS. Outcomes of infants undergoing robot-assisted laparoscopic pyeloplasty compared to open repair. J Urol. 2013 Dec;190(6):2221-6. doi: 10.1016/j.juro.2013.07.063. Epub 2013 Aug 1. PMID 23911637
- [Background] Srougi V, Yorioka M, Sanchez DC, Onal B, Houck CS, Nguyen HT. The feasibility of robotic urologic surgery in infants and toddlers. J Pediatr Urol. 2013 Dec;9(6 Pt B):1198-203. doi: 10.1016/j.jpurol.2013.05.011. Epub 2013 Jun 17. PMID 23782875
- [Background] Yee DS, Shanberg AM, Duel BP, Rodriguez E, Eichel L, Rajpoot D. Initial comparison of robotic-assisted laparoscopic versus open pyeloplasty in children. Urology. 2006 Mar;67(3):599-602. doi: 10.1016/j.urology.2005.09.021. Epub 2006 Feb 28. PMID 16504272
- [Background] Greenfield S, Kaplan SH. Building useful evidence: changing the clinical research paradigm to account for comparative effectiveness research. J Comp Eff Res. 2012 May;1(3):263-70. doi: 10.2217/CER.12.23. PMID 23577230
- [Background] Sequist TD, Schneider EC, Anastario M, Odigie EG, Marshall R, Rogers WH, Safran DG. Quality monitoring of physicians: linking patients' experiences of care to clinical quality and outcomes. J Gen Intern Med. 2008 Nov;23(11):1784-90. doi: 10.1007/s11606-008-0760-4. Epub 2008 Aug 28. PMID 18752026
- [Background] Freilich DA, Penna FJ, Nelson CP, Retik AB, Nguyen HT. Parental satisfaction after open versus robot assisted laparoscopic pyeloplasty: results from modified Glasgow Children's Benefit Inventory Survey. J Urol. 2010 Feb;183(2):704-8. doi: 10.1016/j.juro.2009.10.040. Epub 2009 Dec 21. PMID 20022046
- [Background] Ostlie DJ, St Peter SD. The current state of evidence-based pediatric surgery. J Pediatr Surg. 2010 Oct;45(10):1940-6. doi: 10.1016/j.jpedsurg.2010.05.008. PMID 20920710
- [Background] Chapman SJ, Shelton B, Mahmood H, Fitzgerald JE, Harrison EM, Bhangu A. Discontinuation and non-publication of surgical randomised controlled trials: observational study. BMJ. 2014 Dec 9;349:g6870. doi: 10.1136/bmj.g6870. PMID 25491195
- [Background] Sanematsu H, Wiehe SE. Insight 2: Engaging the health humanities. 2013
- [Background] Sanematsu H, Wiehe S. Learning to look: Design in health services research. Touchpoint 2014
- [Background] Abraham NS, Hewett P, Young JM, Solomon MJ. Non-entry of eligible patients into the Australasian Laparoscopic Colon Cancer Study. ANZ J Surg. 2006 Sep;76(9):825-9. doi: 10.1111/j.1445-2197.2006.03878.x. PMID 16922907
- [Background] Jorgensen LN, Rosenberg J, Al-Tayar H, Assaadzadeh S, Helgstrand F, Bisgaard T. Randomized clinical trial of single- versus multi-incision laparoscopic cholecystectomy. Br J Surg. 2014 Mar;101(4):347-55. doi: 10.1002/bjs.9393. PMID 24536008
- [Background] Sanematsu H, Hong Y, Cole L. Listening through Seeing: Using Design Methods to Learn about the Health Perceptions of Garden on the Go Customors. Indianapolis: 2014
- [Background] Bennet A, Eglash R, Krishnamoorthy M, Rarieya M. Audience as Co-Designer: Participatory Design of HIV/AIDS Awareness & Prevention Posters in Kenya. In: Design Studies. New York: 2006. p. 179-97
- [Background] Sanematsu H. 53. Fun with Facebook: The Impact of Focus Groups on the Development of Awareness Campaigns for Adolescent Health. Journal of Adolescent Health 2011;48(2):S44-5
- [Background] Bate P, Robert G. Experience-based design: from redesigning the system around the patient to co-designing services with the patient. Qual Saf Health Care. 2006 Oct;15(5):307-10. doi: 10.1136/qshc.2005.016527. PMID 17074863
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Durani P, McGrouther DA, Ferguson MW. The Patient Scar Assessment Questionnaire: a reliable and valid patient-reported outcomes measure for linear scars. Plast Reconstr Surg. 2009 May;123(5):1481-1489. doi: 10.1097/PRS.0b013e3181a205de. PMID 19407619

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic Surgery | Open Surgery
Started | 5 | 6
1 Week Post op | 5 | 6
2 Week Post op | 4 | 6
6 Week Post op | 4 | 6
3 Month Follow up (Timing is 3 months after the 6 week post op visit) | 4 | 5
Completed | 4 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic Surgery | Open Surgery | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Customized [Count of Participants; unit: Participants]
  Age 2 to 8 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Length of Post Op Inpatient Hospital Stay Measured in Days
Description: Number of inpatient hospital days post surgery obtained via retrospective chart.
Time Frame: surgery to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 5 | 6
days | 1 (0) | 1 (0)

2. Primary Outcome: Number of Doses of Narcotic Pain Medication In the First 24 Hours Post Op
Description: Pain medication use during hospitalization obtained via retrospective chart review. Dose recorded in mg and frequency recorded as number of doses administered in 24 hour period
Time Frame: Surgery to the first 24 hours post op
Measure: Mean (Standard Deviation); unit: Number of Doses
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 5 | 6
Number of Doses | 0.600 (0.550) | 0.500 (0.550)

3. Primary Outcome: Total Dose of Narcotic Pain Medication In the First 24 Hours Post Op in Morphine Milligram Equivalents (MME)
Description: Pain medication use during hospitalization obtained via retrospective chart review. Morphine milligram equivalents (MME) are values that represent the potency of an opioid dose relative to morphine
Time Frame: Surgery to the first 24 hours post op
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 5 | 6
MME | 1.2 (1.10) | 0.500 (0.550)

4. Primary Outcome: Grade of Surgical Complications up to 1 Year Post op Using Clavian-Dindo Classification
Description: This s a standardized scale to rank the severity of a surgical complication. The higher the grade the more severe the surgical complication. Minimum value is Grade "0" no complication to maximum Grade IV life threatening complication. Grades I thru IV defined as:
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.
  This grade also includes wound infections opened at the bedside ; Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusionsand total parenteral nutritionare also included; Grade III Requiring surgical, endoscopic or radiological intervention; Grade IV Life-threatening complication (including CNS complications)* requiring IC/ICU-management
Time Frame: up to 1 year post up
Measure: Mean (Standard Deviation); unit: grade on a scale
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 5 | 6
grade on a scale | 0.6 (1.34) | 0 (0)

5. Primary Outcome: Pain Score Measured Using The FLACC at 2 Week Post Op Follow Up
Description: Obtained from hospital record and participant report post discharge via the FLACC (behavioral scale for scoring postoperative pain in young children). FLACC score range: minimum "0" ( comfortable) and "10" (severe discomfort)
Time Frame: 1 week post op follow up
Population: FLACC scores 2 week post op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 4 | 5
score on a scale | 2.5 (3.70) | 0 (0)

6. Primary Outcome: Length Of Time For Patient To Return To Normal Routine After Surgery Measured in Days at 2 Week Post Follow Up
Description: Study team created a questionnaire to better understand patient's post op experience. Participant to complete questionnaire with targeted questions on: Side effects of medication and impact; Experience of having a temporary ureteral stent; Ease of removing stent; Return to activity; Financial burden reported by family. No scale or scoring utilized to assess outcome.
Time Frame: 2 week post op follow up
Population: Participant asked "At this point in your child's post op recovery, has your home routine returned to normal?" If participant responded "Yes" then participant asked "Estimate the length of time length of time it took to return to normal."
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 3 | 6
days | 7.67 (5.03) | 6.5 (3.73)

7. Primary Outcome: Length Of Time Parent Was Out Of Work After Child's Surgery Measured in Days at 2 Week Post Follow Up
Description: Number of days parent out of work after operation obtained by parent report. No scale or scoring utilized to assess outcome.
  Participant asked "Have you returned to work since your child's surgery?". If "Yes", asked to estimate the length of time you were out of work after your child's operation.
Time Frame: 2 week post op follow up
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 3 | 4
days | 3.33 (3.51) | 5 (3.92)

8. Primary Outcome: Satisfaction With Scar Appearance Measured Using the Patient Scar Assessment Questionnaire at 3 Month Follow Up Visit
Description: Participant completed the Patient Scar Assessment Questionnaire (PSAQ) at 3 month follow up visit. The 3 month follow up was scheduled at the 6 week post op visit. The "Satisfaction with Appearance" subscale consists of a 8 items with 4-point categorical responses, scoring 1 to 4 points (with 1 point assigned to the most favourable category and 4 assigned to the least favourable). The minimum score of this scale is an "8" and maximum "32."
Time Frame: up to 3 month follow up visit (18 weeks post op)
Population: Satisfaction with Appearance at 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 4 | 5
score on a scale | 10.25 (3.86) | 11.40 (3.05)

9. Primary Outcome: Satisfaction With Symptoms Measured Using the Patient Scar Assessment Questionnaire at 3 Month Follow Up Visit
Description: The Patient Scar Assessment Questionnaire (PSAQ) was completed at the 3 month follow up (scheduled at the 6 week post op visit).
  Higher scores reflect a poorer perception of the scar related to the domain being evaluated. The "Satisfaction with Symptoms" subscale consists of a 5 items with 4-point categorical responses, scoring 1 to 4 points (with 1 point assigned to the most favourable category and 4 assigned to the least favourable). The minimum score of this scale is an "5" and maximum "20.
Time Frame: up to 3 month follow up visit (18 weeks post op)
Population: Satisfaction with Appearance at 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 4 | 5
score on a scale | 5.50 (1) | 7 (2.74)

10. Primary Outcome: Quality of Life Measured Using The Glasgow Children's Benefit Inventory at 3 Month Follow Up Visit
Description: Participant completed the GCBI at 3 month follow up visit. The 3 month follow up was scheduled at the 6 week post op visit.
  The Glasgow Children's Benefit Inventory (GCBI). is a 24 question 5 point Likert scale 2 (much better) to -2 (much worse) with scoring range from -100 (maximum harm) to +100 (maximum benefit).
Time Frame: 3 month follow up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Robotic Surgery | Open Surgery
Number analyzed (Participants) | 4 | 5
score on a scale | 14.08 (32.42) | 20.88 (31.86)

ADVERSE EVENTS:
Time Frame: 3yr 8 months
Description: Study start (10.24.17) to Study end (6.23.21)
Arm/Group | Robotic Surgery | Open Surgery
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04884945/Prot_001.pdf